CLINICAL TRIAL: NCT06657859
Title: A Phase 2, Open-Label Extension Study to Assess the Safety and Efficacy of GLM101 Administered Intravenously to Participants With PMM2-CDG
Brief Title: Open-Label Extension Study to Assess GLM101 in PMM2-CDG Patients
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Glycomine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLM101-007
Record Dates: First submitted 2024-10-22; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Pmm2-CDG; Phosphomannomutase 2 Deficiency
Keywords: GLM101; Pmm2; CDG; CDG 1a
MeSH Terms: conditions — Congenital disorder of glycosylation type 1A

STUDY DESIGN:
Intervention Model Description: This is an open-label extension study. Participants will continue to receive the same dose level they received in the prior study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 10 mg/kg GLM101 (Experimental): GLM101 IV infusions, given weekly
  Interventions: Drug: GLM101
- 20 mg/kg GLM101 (Experimental): GLM101 IV infusions, given weekly
  Interventions: Drug: GLM101
- 30 mg/kg GLM101 (Experimental): GLM101 IV infusions, given weekly
  Interventions: Drug: GLM101

INTERVENTIONS:
Drug: GLM101 — GLM101 IV infusion

SUMMARY:
The goal of this clinical trial is to provide continued access to GLM101 to treat PMM2-CDG in people who have previously received GLM101 in other trials. It will also learn about the long term safety of GLM101. Participants will complete weekly infusions of GLM101 at the same dose level received in previous trials.

DETAILED DESCRIPTION:
This is a phase 2 open-label clinical study of GLM101 in patients with PMM2-CDG who have previously participated in a study of GLM101. This study is designed to monitor long-term safety and treatment effect of GLM101 and provided continued access to study treatment. Participants will continue weekly infusions of GLM101 at the same dose level they received in the previous study. Dose levels may be adjusted to lower doses or higher doses based on available data that demonstrates a change to be safe and tolerable. Participants will be asked to complete questionnaires to evaluate changes in ataxia and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent/assent and/or their legally authorized representative
* Completed previous clinical study with GLM101
* If female of childbearing potential, must not be pregnant and use a medically accepted method of contraception
* If male and sexually active must agree to use a medically acceptable method of contraception
* Willing ad able to adhere to study requirements described in the protocol

Exclusion Criteria:

* Has a condition that would compromise safety or compliance of participant or preclude participant completion of study
* Has positive serum pregnancy test
* Unwilling or unable to comply with scheduled visits, study drug administration plan, laboratory tests, other study procedures, and study restrictions.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate long-term safety | From enrollment to end of treatment up to 4 years
  Number of participants with treatment related adverse events as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

SECONDARY OUTCOMES:
Evaluate changes in ataxia using International Cooperative Ataxia Rating Scale (ICARS) | From enrollment, at 3 months, 6 months and annually to end of treatment up to 4 years
  The scale is scored out of 100 with 19 items and 4 subscales of postural and gait disturbances, limb ataxia, dysarthria, and oculomotor disorders. Higher scores indicate higher levels of impairment.
Maximum observed plasma concentration (Cmax) | From enrollment to end of treatment up to 4 years
  Assessment of the pharmacokinetics (PK) of GLM101
Time to maximum observed plasma concentration (Tmax) | From enrollment to end of treatment up to 4 years
  Assessment pharmacokinetics (PK) of GLM101
Area under the plasma concentration vs. time curve (AUC) | From enrollment to end of treatment up to 4 years
  Assessment of the pharmacokinetics (PK) of GLM101

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Glycomine, Inc.
Locations (1):
- Hospital Sant Joan de Déu, Barcelona, Spain